CLINICAL TRIAL: NCT01533844
Title: An Observational, Non-interventional Study to Determine the Role of Clostridium Difficile in the Pathogenesis of Disease Observed in Neonates and to Investigate the Feasibility of a Potential Study to Evaluate Safety, Efficacy and Pharmacokinetics of Fidaxomicin Oral Suspension in Neonates With Clostridium Difficile Associated Disease (CDAD)
Brief Title: To Determine the Feasibility of a Fidaxomicin Study in Neonates and to Assess C. Difficile (Clostridium Difficile) Involvement in the Pathogenesis
Acronym: DAISY
Status: Terminated | Type: Observational
Why Stopped: Terminated due to the fact that the required number of trial subjects was not met.
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 2819-CL-0204
Record Dates: First submitted 2012-02-13; First posted 2012-02-15 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Clostridium Difficile
Keywords: CDAD; Neonates; Clostridium difficile

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool Sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neonates: Neonates with CDAD

SUMMARY:
The objective of this multi-center, prospective observational study is to determine the feasibility of a potential interventional study with fidaxomicin. The incidence and clinical aspects of Clostridium difficile infection (CDI) in neonates will be determined, and it will be assessed whether a subgroup can be identified where treatment with fidaxomicin therapy might improve outcome.

ELIGIBILITY:
Inclusion Criteria:

* Subject is suffering from diarrhea or other signs or symptoms consistent with CDAD (as described in section 5.2.3)
* Presence of either toxin A or B (or both) of C. difficile in the stool within 24 hours prior to enrollment using the C. difficile Quik Chek Complete® diagnostic test, provided by the sponsor

Exclusion Criteria:

Subject will be excluded from participation if any of the following apply:

* Preterm neonates
* Negative C. difficile toxin test

Max Age: 27 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Term neonates less than 28 days of age at enrollment, referred to healthcare professionals due to suspected C Difficile Associated Disease (CDAD).
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of a potential interventional study with fidaxomicin | 40 days
  The incidence and clinical aspects of clostridium difficile infection (CDI) in neonates will be determined, and it will be assessed whether a subgroup can be identified where treatment with fidaxomicin therapy might improve outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (9):
- France (2):
  - Site: 3301, Poissy, Paris
  - Site: 3302, Lyon
- Germany (3):
  - Site: 4902, Erlangen
  - Site: 4904, Hanover
  - Site: 4901, Munich
- Site: 3102, Maastricht, Netherlands
- Spain (3):
  - Site: 3403, Granada
  - Site: 3402, Madrid
  - Site: 3401, Valencia